CLINICAL TRIAL: NCT06172452
Title: Testing a Single-Session Online Body Image and Mood Program for Sexual and Gender Minority (SGM) Adolescents
Brief Title: Randomized Controlled Trial of Project Body Neutrality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jessica Schleider, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00220039
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-02

CONDITIONS: Depression; Eating Disorders; Body Image
MeSH Terms: conditions — Depression; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the intervention condition or the supportive therapy control.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Project Body Neutrality SSI (Experimental): Project Body Neutrality is a digital, self-guided SSI that teaches adolescents about body neutrality. It contains self-reflection exercises, vignettes from fictional peers, and psychoeducation that support users in understanding why body positivity may be a difficult mindset for some individuals to obtain; additional self-reflection exercises and vignettes that present body neutrality as a well-rounded alternative to body positivity; exercises that culminate in a user-generated list of activities that their body allows them to enjoy as well as statements they can use to counter negative thoughts about their body; writing prompts where users provide advice based on body neutrality principles to fictional peers struggling with their body image; and an opportunity to contribute their advice or reflections anonymously to a lab-run social media campaign as a form of body neutrality advocacy. See all materials for this intervention here: https://osf.io/7qtuj.
  Interventions: Behavioral: Project Body Neutrality SSI
- Supportive Therapy SSI (Placebo Comparator): The Sharing Feelings SSI is a digital, self-guided SSI that is structurally similar to Project Body Neutrality, but it is designed to mimic supportive therapy (ST). The goals of the ST intervention are to encourage participants to identify and express feelings to close others; the intervention does not teach or emphasize specific skills or beliefs. The ST-SSI is designed to control for nonspecific aspects of intervention, including engagement in a computer program, reading and writing exercises, and vignettes from fictional peers. See all materials for this intervention here: https://osf.io/u4axs/.
  Interventions: Behavioral: Supportive Therapy SSI

INTERVENTIONS:
Behavioral: Project Body Neutrality SSI — Online, 30-minute self-guided intervention for youth ages 13-17
  Arms: Project Body Neutrality SSI
Behavioral: Supportive Therapy SSI — Online, 30-minute self-guided activity for youth ages 13-17
  Arms: Supportive Therapy SSI

SUMMARY:
This study tests a single-session intervention (SSI) targeting risk factors for depression and eating disorders among sexual and gender minority (SGM) adolescents. Youth ages 13-17 who identify as sexual or gender minorities will be randomized to the intervention condition (Project Body Neutrality SSI) or a control (supportive therapy SSI). Participants will complete questionnaires before the intervention, immediately after the intervention, and 3-months after completing the intervention so that the study team can investigate if Project Body Neutrality leads to reductions in depression and eating disorder symptoms compared to the control.

ELIGIBILITY:
Inclusion Criteria:

* Identify as a sexual or gender minority individual per self-report
* 13-17 years old at the time of enrollment
* English proficiency per self-report
* Report having body image concerns per self-report
* Score of ≥ 2 on the Patient Health Questionnaire-2 (PHQ-2; Kroenke et al., 2003), - indicating elevated depressive symptoms
* Did not participate in a past study involving Project Body Neutrality per self-report
* Residing within the United States per IP address
* Passes comprehension of consent language assessment

Exclusion Criteria:

* Fail to meet the above-listed inclusion criteria
* Exit the study prior to condition randomization
* Failure to pass the data integrity measures
* Duplicate responses from the same individual in baseline or follow-up surveys

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Examination Questionnaire - 10 item, 3 factor version (EDE-Q; Fairburn & Beglin, 2008; Habashy et al., 2023) | Pre-Intervention to 3-month follow-up
  A 10-item questionnaire designed to assess the range and severity of features associated with a diagnosis of eating disorder. The original measure's factor structure has failed to replicate across many samples, especially for diverse populations. This version has achieved strict invariance by gender and race/ethnicity. Higher global scores indicate greater eating disorder severity (primary outcome). Outcomes for the three subscales (Dietary Restaurant, Preoccupation with Eating Concern, and Shape/Weight Overvaluation) will also be reported. Each item is on a 0 to 6 scale and the scores are computed as means.
Short Mood and Feelings Questionnaire (SMFQ; Messer et al., 1995) | Pre-Intervention to 3-month follow-up
  A 13-item questionnaire designed to assess depressive symptoms in youth. Total scores range from 0 to 26, with higher scores indicating greater depression severity (primary outcome).

SECONDARY OUTCOMES:
Beck Hopelessness Scale - 4 item version (BHS; Perczel Forintos et al., 2013) | Pre-Intervention to Immediately Post-Intervention; Pre-Intervention to 3-month follow-up
  Asks respondents to rate four statements reflecting their sense of hopelessness from 0 (Absolutely Disagree) to 3 (Absolutely Agree). Total scores range from 0 to 12, with higher scores indicating greater levels of hopelessness.
State Hope Scale - 3 item Pathways subscale (SHS; Snyder et al., 1996) | Pre-Intervention to Immediately Post-Intervention; Pre-Intervention to 3-month follow-up
  Asks respondents to rate three statements from 1 (Definitely False) to 8 (Definitely True). Total score ranges from 3 to 24, with higher scores reflecting greater perceived ability to identify goal-oriented routes.
Functionality Appreciation Scale (FAS; Alleva et al., 2017) | Pre-Intervention to Immediately Post-Intervention; Pre-Intervention to 3-month follow-up
  Asks respondents to rate seven statements from 1 (Strongly Disagree) to 5 (Strongly Agree). Total scores range from 7 to 35, where higher scores indicate greater appreciation for body functionality.
Body Image States Scale (BISS; Cash et al., 2002) | Pre-Intervention to Immediately Post-Intervention; Pre-Intervention to 3-month follow-up
  Asks respondents to rate six items from 1 (poor body image state) to 9 (favorable body image state). Total scores range from 6 to 54, where higher scores indicate a more favorable body image state.

OTHER OUTCOMES:
Body Image Acceptance and Action Questionnaire (BI-AAQ; Sandoz et al., 2013) | Pre-Intervention to Immediately Post-Intervention; Pre-Intervention to 3-month follow-up
  Asks respondents to rate twelve items from 1 (Never True) to 7 (Always True). Total scores range from 12 to 84, with higher scores indicating greater body image flexibility.
Comprehensive Inventory of Mindfulness Experiences for Adolescents - Accepting with Nonjudgmental Orientation Subscale (CHIME-A; Johnson et al., 2017) | Pre-Intervention to Immediately Post-Intervention; Pre-Intervention to 3-month follow-up
  Asks respondents to rate three items from 1 (Almost Never) to 6 (Almost Always). Total scores range from 3 to 18 with higher scores indicating greater nonjudgmental acceptance. We adapted the items of this subscale to ask specifically about nonjudgmental acceptance of one's physical appearance.
Muscle Dysmorphic Disorder Inventory (MDDI; Hildebrandt et al., 2004) | Pre-Intervention to 3-month follow-up
  Asks respondents to rate thirteen items from 1 (Never) to 5 (Always). Total scores range from 13 to 65 with higher scores reflecting a greater severity of muscle dysphoria symptoms.
Program Feedback Scale (PFS; Schleider et al., 2019) | Immediately Post-Intervention
  Asks respondents to rate seven statements regarding intervention acceptability and feasibility; it also includes open-ended items that invite respondents to share what they liked and/or would change about the intervention. The seven statements are rated from 1 (Really Disagree) to 5 (Really Agree). Total score ranges from 5 to 35, with higher scores indicating a more positive evaluation.
Treatment seeking questions | 3-month follow-up
  Respondents are asked two questions about mental health treatment seeking in the past three months: "In the past 3 months (since completing the first survey for this study), did you seek out any new support for depression or mood problems?" and "In the past 3 months (since completing the first survey for this study), did you seek out any new support for an eating disorder or body image problems?"

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Schleider, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alleva JM, Tylka TL, Kroon Van Diest AM. The Functionality Appreciation Scale (FAS): Development and psychometric evaluation in U.S. community women and men. Body Image. 2017 Dec;23:28-44. doi: 10.1016/j.bodyim.2017.07.008. Epub 2017 Aug 17. PMID 28822275
- [Background] Cash TF, Fleming EC, Alindogan J, Steadman L, Whitehead A. Beyond body image as a trait: the development and validation of the Body Image States Scale. Eat Disord. 2002 Summer;10(2):103-13. doi: 10.1080/10640260290081678. PMID 16864251
- [Background] Fairburn CG, Beglin SJ. Eating disorder examination questionnaire. Cognitive Behavior Therapy and Eating Disorders. 2008; 309: 313.
- [Background] Habashy J, Benning SD, Renn BN, Borgogna NC, Lawrence EM, Kraus SW. Psychometric properties of the eating disorder examination questionnaire: Factor analysis and measurement invariance by race/ethnicity and gender. Eat Behav. 2023 Jan;48:101696. doi: 10.1016/j.eatbeh.2022.101696. Epub 2022 Dec 7. PMID 36516727
- [Background] Hildebrandt T, Langenbucher J, Schlundt DG. Muscularity concerns among men: development of attitudinal and perceptual measures. Body Image. 2004 May;1(2):169-81. doi: 10.1016/j.bodyim.2004.01.001. PMID 18089149
- [Background] Johnson C, Burke C, Brinkman S, Wade T. Development and validation of a multifactor mindfulness scale in youth: The Comprehensive Inventory of Mindfulness Experiences-Adolescents (CHIME-A). Psychol Assess. 2017 Mar;29(3):264-281. doi: 10.1037/pas0000342. Epub 2016 Jun 2. PMID 27254018
- [Background] Kroenke K, Spitzer RL, Williams JB. The Patient Health Questionnaire-2: validity of a two-item depression screener. Med Care. 2003 Nov;41(11):1284-92. doi: 10.1097/01.MLR.0000093487.78664.3C. PMID 14583691
- [Background] Messer SC, Angold A, Costello EJ, Loeber R, Van Kammen W, Stouthamer-Loeber M. Development of a short questionnaire for use in epidemiological studies of depression in children and adolescents: Factor composition and structure across development. International Journal of Methods in Psychiatric Research. 1995; 5: 251-262.
- [Background] Perczel Forintos D, Rozsa S, Pilling J, Kopp M. Proposal for a short version of the Beck Hopelessness Scale based on a national representative survey in Hungary. Community Ment Health J. 2013 Dec;49(6):822-30. doi: 10.1007/s10597-013-9619-1. Epub 2013 Jun 12. PMID 23756722
- [Background] Sandoz EK, Wilson KG, Merwin RM, Kate Kellum, K. Assessment of body image flexibility: The Body Image-Acceptance and Action Questionnaire. Journal of Contextual Behavioral Science. 2013; 2(1): 39-48.
- [Background] Schleider JL, Mullarkey MC, Weisz JR. Virtual Reality and Web-Based Growth Mindset Interventions for Adolescent Depression: Protocol for a Three-Arm Randomized Trial. JMIR Res Protoc. 2019 Jul 9;8(7):e13368. doi: 10.2196/13368. PMID 31290406
- [Background] Snyder CR, Sympson SC, Ybasco FC, Borders TF, Babyak MA, Higgins RL. Development and validation of the State Hope Scale. J Pers Soc Psychol. 1996 Feb;70(2):321-35. doi: 10.1037//0022-3514.70.2.321. PMID 8636885
- [Derived] Smith AC, Ahuvia IL, Zapata JP, Cohen KA, Graham AK, Schleider JL. Randomized trial of a digital single-session intervention for body image and mood concerns among LGBTQ+ adolescents. Behav Res Ther. 2025 Oct;193:104809. doi: 10.1016/j.brat.2025.104809. Epub 2025 Jun 24. PMID 40578276